CLINICAL TRIAL: NCT00878774
Title: An Escalating, Multiple-dose Study in Ragweed Allergic Subjects to Assess the Safety of Intradermal Injection of ToleroMune Ragweed
Brief Title: Safety of ToleroMune Ragweed to Treat Ragweed Allergy in Ragweed Allergic Subjects With Rhinoconjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry)
Responsible Party: Dr Rod Hafner, Circassia Limited
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TR001
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-11

CONDITIONS: Allergy
Keywords: Ragweed allergy; Immunotherapy; Rhinoconjunctivitis; Toleromune Ragweed
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): ToleroMune Ragweed, subjects to receive either active or placebo comparator
  Interventions: Biological: ToleroMune Ragweed; Biological: Placebo
- Cohort 2 (Experimental): ToleroMune Ragweed or placebo comparator
  Interventions: Biological: ToleroMune Ragweed; Biological: Placebo
- Cohort 3 (Experimental): ToleroMune Ragweed or placebo comparator
  Interventions: Biological: ToleroMune Ragweed; Biological: Placebo
- Cohort 4 (Experimental): ToleroMune Ragweed or placebo comparator
  Interventions: Biological: ToleroMune Ragweed; Biological: Placebo
- Cohort 5 (Experimental): ToleroMune Ragweed or placebo comparator
  Interventions: Biological: ToleroMune Ragweed; Biological: Placebo

INTERVENTIONS:
Biological: ToleroMune Ragweed — ToleroMune Ragweed dose 1x4 administrations 2 weeks apart
Biological: Placebo — Placebo comparator, 1x4 administrations 2 weeks apart

SUMMARY:
It is estimated that 36 million Americans suffer from seasonal allergies and that ragweed is the primary cause of autumn allergies, 87% of patients with ragweed allergy suffer rhinoconjunctivitis. ToleroMune Ragweed is a novel, synthetic, allergen-derived peptide desensitising vaccine, currently being developed for the treatment of ragweed allergy.

The purpose of the present study is to evaluate the safety and tolerability of multiple ascending doses of ToleroMune Ragweed in subjects in subjects with a documented history of allergic rhinoconjunctivitis on exposure to ragweed pollen. The efficacy of ToleroMune Ragweed will also be explored in these subjects using the Late Phase Skin Response, Early Phase Skin Response and Conjunctival Provocation Test.

DETAILED DESCRIPTION:
This study is designed as a randomised, double-blind, placebo-controlled study to evaluate the safety and tolerability of escalating multiple doses of ToleroMune Ragweed in subjects with a documented history of allergic rhinoconjunctivitis on exposure to ragweed pollen. The efficacy of ToleroMune Ragweed will also be explored in these subjects using the LPSR, EPSR, CPT and levels of ragweed specific IgE. A single centre will be initiated first, with a second centre included as a backup, if needed, to enable recruitment numbers to be met.

The study will consist of 3 study periods. In Period 1, Screening will be performed up to a maximum of 8 weeks before randomisation and may consist of one or two visits to the clinic, at the Investigator's discretion. Baseline Challenge will consist of a single visit 1 to 4 weeks before randomisation.

Period 2 (Treatment Period) will consist of 4 visits (Visits 3A-3D) two weeks apart (14±2 days). Subjects who comply with the inclusion/exclusion criteria will be assigned to one of 5 dose groups. The first dose group will receive 4 administrations of ToleroMune Ragweed. Successive dose groups will increasing doses given as 4 administrations of ToleroMune Ragweed, provided the first administration of the previous dose was safe and well tolerated.

In Period 3, Post-treatment Challenge will take place 19-25 weeks after the first administration in the Treatment Period and will be timed to be outside the Ragweed season. However in the event that the Ragweed season lasts beyond 26th October 2009, the PTC will take place 22-28 weeks after the first administration in the Treatment Period. Assessments performed will be identical to those at the Baseline Challenge. Follow-up will be conducted 3-10 days after PTC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years
* A reliable, documented history of rhinoconjunctivitis (sneezing, rhinorrhoea, nasal blockage, itchy/red/sore/watering eyes) on exposure to ragweed for at least 2 years
* Allergy to ragweed, defined by positive skin prick test at the Screening Visit
* LPSR to ragweed allergen 8 hours after intradermal injection of greater than 25mm diameter response
* Positive CPT to ragweed allergen with a score ≥4
* Willing and able to provide written informed consent
* Subjects who are normally active and otherwise judged to be in good health
* The subject must be willing and able to comply with the study requirements
* If the subject is female and of childbearing potential she must practice an acceptable form of contraception, and produce a negative urine pregnancy test on the Screening Visit. A female subject may be included without a negative urine pregnancy test if she can document that she is surgically sterile or at least 2 years post-menopausal

Exclusion Criteria:

* Subjects with an FEV1 <80% of normal
* Subjects who suffer from other seasonal allergies, and cannot complete the clinical study outside the pollen season or are symptomatic for significant perennial rhinitis
* A history of anaphylaxis to ragweed allergen; subjects who have a history of severe drug allergy, angioedema or anaphylactic reactions to food
* Subjects with a history of asthma
* Subjects who have auto-immune or rheumatoid diseases
* Clinical history of immunodeficiency, including immunosuppressant therapy
* Subjects in whom tyrosine metabolism is disturbed
* Current diagnosis of chickenpox or measles or exposure in the last 3 weeks
* Active or quiescent tuberculous infection of the respiratory tract, untreated local or systemic fungal or bacterial or systemic viral infections or parasitic or ocular herpes simplex
* Have symptoms of a clinically relevant illness, in the Investigator's opinion, within 6 weeks prior to Screening Visit
* Allergen immunotherapy during the last 5 years or ragweed immunotherapy ever.
* Subjects who have completed or are undergoing ongoing treatment with anti-IgE-antibody
* Use of the therapies listed in Section 5.9.2 at any time during the study will make the subject ineligible for the study
* Subjects for whom administration of adrenaline is contra-indicated (e.g. subjects with acute or chronic symptomatic coronary heart disease or severe hypertension)
* Subjects being treated with beta-blockers
* The subject has unacceptable symptoms in the 3 days without loratadine prior to the screening visit
* Female subjects who are pregnant, lactating or planning a pregnancy during the study
* Have any clinically relevant abnormalities detected on physical examination
* 12-lead ECG or vital signs (blood pressure, pulse rate, respiratory rate and oral temperature) that are outside normal limits, unless the abnormality is considered not to be of clinical relevance by the Investigator
* Laboratory values (haematology, biochemistry, urine tests) that are outside the normal ranges, unless the abnormality is considered not to be of clinical relevance by the Investigator
* Significant history of alcohol or drug abuse
* History of immunopathological disease
* Positive test for hepatitis B, hepatitis C or HIV at screening
* Have previously been randomised into this study
* Planned travel outside the study area for a substantial portion of the study period
* Have received treatment with an investigational drug within 6 months prior to study screening or have participated in a study with a new formulation of a marketed drug one month prior to study screening
* Have any significant disease or disorder (e.g. cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment) which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results of the study, or the subject's ability to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple intradermal injections of ToleroMune Ragweed in ragweed allergic subjects with allergic rhinoconjunctivitis | 28 weeks

SECONDARY OUTCOMES:
Mean change from baseline in area of the LPSR 8 hours after intradermal challenge with whole ragweed allergen at PTC after ToleroMune Ragweed injection compared to placebo | 28 weeks
Mean change from baseline in area of the EPSR 15 minutes after intradermal challenge with whole ragweed allergen at PTC after ToleroMune Ragweed injection compared to placebo | 28 weeks
Mean change from baseline in CPT score at PTC after ToleroMune Ragweed injection compared to placebo | 28 weeks
Mean change from baseline in concentration of ragweed specific IgE at PTC after ToleroMune Ragweed injection compared to placebo | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Hebert, MD, Principal Investigator — Centre de Recherche Appliqué en Allergie de Québec
Locations (1):
- Centre de Recherche Appliqué en Allergie de Québec, Québec, Quebec, Canada